CLINICAL TRIAL: NCT02283060
Title: Change in Sleep Architecture and Neuropsychological Performance Following Switch From Atripla to Stribild.
Brief Title: Sleep and Cognition After Atripla to Stribild Switch
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Hawaii (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H027
Record Dates: First submitted 2014-10-29; First posted 2014-11-05 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: HIV
Keywords: Atripla; Stribild; HIV; Sleep architecture; Neuropsychological performance
MeSH Terms: interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stribild switch arm (Experimental): Patient to be taken off Atripla and switched to Stribild (co-formulated elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate) -one tablet taken daily with food
  Interventions: Drug: Stribild
- Atripla control arm (Active Comparator): Patient to continue taking Atripla (co-formulated efavirenz/emtricitabine/ tenofovir disoproxil fumarate) - one tablet taken daily at bedtime on an empty stomach
  Interventions: Drug: Atripla

INTERVENTIONS:
Drug: Stribild — To be administered orally, once daily with food.
  Other Names: Co-formulated elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate
  Arms: Stribild switch arm
Drug: Atripla — To be administered orally, once daily at bedtime on an empty stomach
  Other Names: Co-formulated efavirenz/emtricitabine/ tenofovir disoproxil fumarate
  Arms: Atripla control arm

SUMMARY:
Atripla and Stribild are two FDA-Approved one pill a day combination antiretroviral medications given for the treatment of HIV. Both drugs are reasonably well tolerated. However, efavirenz, a component of Atripla, is known to cause "mental" side effects.

This proposal aims to assess whether a switch from Atripla to Stribild for 12 weeks will be associated with reversal of sleep and cognitive disturbances. Demonstrating changes upon withdrawal of drug and substitution of a drug regimen not known to have an impact on sleep and cognition may represent the best option to determine whether use of efavirenz is associated with effects on sleep and cognition beyond the immediate period following initiation of drug.

DETAILED DESCRIPTION:
Atripla (efavirenz/emtricitabine/tenofovir disoproxil fumarate) and Stribild (elvitegravir/emtricitabine/tenofovir disoproxil fumarate/cobicistat) are 2 FDA-approved 'one pill once a day' combination antiretroviral medications given for the treatment of HIV. Both have a common nucleoside reverse transcriptase inhibitor (NRTI) backbone of tenofovir (TDF) and emtricitabine (FTC), but differ in the 3rd medication contained in the pill. Atripla contains a non-nucleoside reverse transcriptase (NNRTI) drug efavirenz (EFV) while Stribild (elvitegravir/emtricitabine/tenofovir disoproxil fumarate/cobicistat) contains an integrase inhibitor elvitegravir with the drug cobicistat inactive against HIV but designed to simply boost the level of elvitegravir.

Both drugs are reasonable well tolerated. However, efavirenz is known to cause 'mental' side-effects. It is known that the initial use of EFV is associated with central nervous system (CNS) toxicity. The symptoms of such toxicity include daytime sleepiness, or alternatively inability to sleep, as well as vivid dreams including nightmares. The majority of such symptoms are believed to resolve within weeks; however there is controversy as to whether residual problems persist on a long term basis. Furthermore there are now reports of long time cognitive dysfunction associated with the use of efavirenz. Whether this is related to sleep disturbance is not clear. Studies to assess this impact have primarily involved assessment of sleep and cognitive function in antiretroviral (ART)-naïve subjects as they are initiated on first time ART that includes EFV. Such studies however are confounded by a 'return to health' phenomena as HIV per se is known to cause sleep and cognitive deficits . There is controversy regarding whether use of efavirenz leads to long term disturbances in sleep and cognition. HIV per se causes sleep and cognitive deficits6 and studies which have tried to assess problems in antiretroviral-naïve subject's pre- and post- initiation of efavirenz-based regimens may be confounded by a 'return to health' phenomena.

This proposal aims to assess whether a switch from efavirenz/emtricitabine/tenofovir disoproxil fumarate to elvitegravir/emtricitabine/tenofovir disoproxil fumarate/cobicistat will be associated with reversal of sleep and cognitive disturbances. Demonstrating changes upon withdrawal of drug and substitution of a drug regimen not known to have an impact on sleep or cognition may represent the best option to determine whether use of EFV is associated with effects on sleep and cognition beyond the immediate period following initiation of drug.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Age 18 to 65 years
* On stable efavirenz/emtricitabine/tenofovir disoproxil fumarate regimen > 12 months
* Documented plasma HIV RNA < 50 copies/ml within 3 months of entry
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Receipt of any other antiretroviral drugs in addition to efavirenz/emtricitabine/tenofovir disoproxil fumarate within 6 months of study entry
* Any documented plasma HIV RNA > 100 copies/ml within the past 6 months prior to study entry
* Chronic hepatitis B as assessed by positive hepatitis B surface antigen [HBsAg]
* Chronic hepatitis C as assessed by positive hepatitis C antibody [HCVab], except with proof of viral clearance and normal liver function tests
* Other chronic disease which is uncontrolled or likely to interfere with study results
* Acute illness within 2 weeks of entry
* Previously documented history of OSA (obstructive sleep apnea)
* Moderate to high risk of OSA defined as BMI (Body mass index) > 30 plus two of the following: habitual snoring, gasping/choking, observed apnea while sleeping, neck circumference > 17 inches
* Severe depression based on the BDI-2 (Beck Depression Inventory - II)
* Chronic daily receipt of medications associated with potential for sleep interference (i.e. psychoactive drugs, steroids, decongestants, beta blockers)
* Any immunomodulator, HIV vaccine, any other vaccine, or investigational therapy within 30 days of study entry.
* Anticipated need for medications which are contraindicated as per Stribild package insert
* Any known contra-indication to use of Stribild (elvitegravir/emtricitabine/tenofovir disoproxil fumarate/cobicistat)
* Creatinine clearance (Cockcroft and Gault) < 70 ml/min
* The following lab values:

  1. Hemoglobin < 9.0
  2. Absolute neutrophil count < 500/μL
  3. Platelet count < 40,000/μL
  4. AST (SGOT) and ALT (SGPT) > 5x ULN
* Active or recent past history (within past 5 years) of illicit substance or alcohol use or abuse which, in the judgment of the Investigator, will interfere with the patient's ability to comply with the protocol requirements
* Pregnancy or breast-feeding, intent to become pregnant during the course of the study or breast-feeding
* Patients, who, in the opinion of the Investigator, are unable to comply with the dosing schedule and protocol evaluation or for whom the study may not be advisable

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change in sleep architecture assessed by formal sleep study | 12 weeks
  Change in sleep architecture as assessed by formal sleep study
Change in neuropsychological performance global and subdomain neuropsychological test scores | 12 weeks
  Change in global and subdomain neuropsychological test scores

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index Score | 12 weeks
Change in the frequency of use of sleep medications | 12 weeks
Change in the quality of life index score | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hawaii Center for AIDS, Honolulu, Hawaii, United States